CLINICAL TRIAL: NCT02965079
Title: Registry on the EXperience of Extracorporeal CO2 Removal in Intensive Care Units
Acronym: REXECOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rexecor (Other)
Responsible Party: Sponsor
Other Study IDs: APHP
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease; Patients With Acute Respiratory Distress Syndrome
Keywords: extracorporeal CO2 removal; registry; COPD and ARDS; CEDIT on behalf of APHP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ECCO2R — The ECCO2R system was developed from the principle of ECMO systems by underscoring the importance of carbon dioxide elimination rather than direct improvement of oxygenation in some patients. The circuit of the ECCO2R system can be set up in venovenous (VV) or arteriovenous (AV). For VV setup, a low flow pump is used to maintain a low extracorporeal flow rate using only 20-30 % of cardiac output. The ECCO2R system does not provide complete pulmonary function as it can achieve only limited oxygenation but provides predominantly carbon dioxide removal. As neither VV nor AV circuit allows full cardiopulmonary bypass, the system provides respiratory function but no cardiac support

SUMMARY:
Investigators will aim to conduct an observational study in order to assess very thoroughly all patients implanted by Extracorporeal carbon dioxide removal (ECCO2R) in 10 critical care units of Paris and its surburb (APHP, Assistance Publique des hôpitaux de Paris).

Secondary objectives will be:

1. to assess efficacy and safety of ECCO2R,
2. to compare the data issue from the registry to others studies assessing the same population and to other centers and
3. to compare the different ECCOR devices in terms of efficacy and adverse events.

DETAILED DESCRIPTION:
The registry will be conducted prospectively during 2 years in 10 ICUs of l'APHP on behalf on the CEDIT. The 10 centers are : (1) ICU of l'hôpital europeén Georges Pompidou, (2) ICU of l'Hôpital Louis Mourier, (3) ICU of l'Hôpital de Bicêtre, (4) ICU of GHPS, (5) Respiratory ICU of GHPS, (6) ICU of l'Hôpital Lariboisière (7) ICU of l'Hôpital Cochin (8) ICU of l'Hôpital Saint-Antoine (9)ICU of l'Hôpital Henri Mondor and (10) ICU of l'Hôpital Tenon.

The primary outcome will be the number of patients implanted by ECCO2R monthly in each center during the 2 years period study.

Secondary outcomes will be ICU-mortality, invasive ventilation duration, non invasive ventilation duration, ICU duration, modalities of ventilation at the ICU discharge, hemorragic complications due to the ECCOR device, thrombotic complications due to ECCO2R device, intravascular hemolysis due to ECCO2R device, duration of ECCO2R, adjunct therapy to ECCO2R and reasons of ECCO2R discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with ECCCO2R

Exclusion Criteria:

* Contra-indication to ECCO2R

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 types of patients : Patients with acute exacerbation of chronic obstructive pulmonary disease (COPD) and acute hypercapnic respiratory failure at high risk to failed noninvasive ventilation Patients with acute exacerbation of chronic obstructive pulmonary disease (COPD) needing invasive ventilation in order to reduce mechanical ventilation duration Patients with ARDS and with the ail to reduce ventilation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of ECCO2R use | Recorded monthly up to 100 weeks (24 months)
  Number of ECCO2R implantation monthly by center

SECONDARY OUTCOMES:
ICU mortality | Recorded From date of ICU admission until the date of death or ICU discharge, assessed up to 100 weeks
Duration of mechanical ventilation | Recorded from ICU admission until the date of death or ICU discharge,assessed up to 100 weeks
ICU duration | Recorded from ICU admission until the date of death or ICU discharge,assessed up to 100 weeks
Ventilation modalities at discharge | Recorded from the initiation of ventilation until ventilation removal,assessed up to 100 weeks
hemorragic and thrombotic complications | Recorded from the date of ECCO2R implantation until the removal of the device,assessed up to 100 weeks
hemolysis | Recorded from the date of ECCO2R implantation until the removal of the device,assessed up to 100 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique - Hopitaux de Paris, Paris, France

REFERENCES:
- [Derived] Augy JL, Aissaoui N, Richard C, Maury E, Fartoukh M, Mekontso-Dessap A, Paulet R, Anguel N, Blayau C, Cohen Y, Chiche JD, Gaudry S, Voicu S, Demoule A, Combes A, Megarbane B, Charpentier E, Haghighat S, Panczer M, Diehl JL. A 2-year multicenter, observational, prospective, cohort study on extracorporeal CO2 removal in a large metropolis area. J Intensive Care. 2019 Aug 20;7:45. doi: 10.1186/s40560-019-0399-8. eCollection 2019. PMID 31452899